CLINICAL TRIAL: NCT00840736
Title: Laparoscopic Adjustable Gastric Banding Versus Open Vertical Banded Gastroplasty: 7-Year Results of a Prospective Randomized Trial
Brief Title: LAGB Versus VBG: 7-Year Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Jan Willem M. Greve, MD PhD, Atrium Medical Centre Parkstad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAGBvsVBG7y
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Morbid Obesity; Bariatric Surgery; Vertical Banded Gastroplasty; Laparoscopic Adjustable Gastric Banding; Long Term Results
Keywords: VBG; LAGB; long term results; Weight loss; Complications; Reoperations; Conversion
MeSH Terms: conditions — Obesity, Morbid; Weight Loss | interventions — Gastroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Laparoscopic adjustable gastric banding
  Interventions: Procedure: Laparoscopic adjustable gastric banding
- 2 (Active Comparator): vertical banded gastroplasty
  Interventions: Procedure: vertical banded gastroplasty

INTERVENTIONS:
Procedure: Laparoscopic adjustable gastric banding — Laparoscopic adjustable gastric banding
  Other Names: LAGB, AGB, LB, lap-band, SAGB
  Arms: 1
Procedure: vertical banded gastroplasty — vertical banded gastroplasty
  Other Names: VBG, Mason, gastroplasty
  Arms: 2

SUMMARY:
The study aims to investigate the long term results of a randomized clinical single-centre trial comparing two standard operative techniques in bariatric surgery; laparoscopic adjustable gastric banding and vertical banded gastroplasty.

DETAILED DESCRIPTION:
One hundred morbidly obese patients were included in the study. Randomization between the two operative techniques was performed using a computer model. Fifty patients were included in both groups. Weight loss, obesity-related comorbidity, long term complications, re-operations and conversions were all prospectively investigated for a mean period of 84 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI of > 40 kg/m2 or > 35 kg/m2 with obesity-related comorbidities
* Failure to achieve sustainable weight loss with proven conservative measures

Exclusion Criteria:

* severe psychiatric and / or eating disorders
* unable to keep to a prescribed postoperative diet
* < 18 or > 60 years
* not eligible to bariatric surgery according to a member of the multidisciplinary team (psychologist, dietician, nurse practitioner, general practitioner and surgeon)

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
weight loss | 84 months

SECONDARY OUTCOMES:
co-morbidity | 84 months
complications | 84 months
reoperations / revisions / conversions | 84 months
Quality of life | 84 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem M Greve, Md PhD, Study Director — Atrium Medical Centre Parkstad; Ruben Schouten, MD, Principal Investigator — Atrium Medical Centre Parkstad
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands